CLINICAL TRIAL: NCT06031909
Title: Multimodal Assessment of Frailty in Acute Stroke Patients Treated at a Certified Stroke-unit
Brief Title: Multimodal Assessment of Frailty in Acute Stroke Patients
Acronym: MAFASP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Stefan Gerner, Principal Investigator, Associate professor, University of Giessen
Other Study IDs: AZ 220/21
Record Dates: First submitted 2023-08-30; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Stroke; Frailty
Keywords: frailty; outcome; elderly
MeSH Terms: conditions — Stroke; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patients: Stroke patients admitted to the certified stroke-unit of the Department of Neurology, University Hospital Giessen, Germany.
  Interventions: Diagnostic Test: Multimodal frailty assessment

INTERVENTIONS:
Diagnostic Test: Multimodal frailty assessment — Different domains are assessed during hospital stay, these include:
  * Clinical scores: Clinical Frailty scale (CFS), Groningen Frailty index (GFI)
  * Brain frailty: assessing white matter hyperintensieties, atrophy and lacunar strokes in initial brain imaging
  * Laboratory values: laboratory Frailty index (FI-Lab), inflammatory markers
  * Nutrition: Controlling nutritional status score (CONUT-score), body mass index, dysphagia assessment (FOIS)
  * Mobility/strengths: de Morton Mobility Index (DEMMI), grip strenghts of non-paralytic arm via dynamometer, muscle mass estimated by sonographic measurement of the biceps brachii muscle and the rectus femoris muscle.

SUMMARY:
The goal of this study is to investigate the influence of frailty on clinical and stroke characteristics, treatment and outcomes in patients with acute stroke.

The main questions it aims to answer are:

1. How prevalent is frailty in patients with stroke?
2. Which impairments (e.g. undernutrion, impaired mobility, laboratory markers) contribute to frailty?
3. Is the outcome of frail patients worse than those without?
4. Are in-hospital complications more frequent in frail patients than those without?

DETAILED DESCRIPTION:
Stroke is one of the most common causes of disability and mortality worldwide. A recognized complication in stroke patients is frailty, which is associated with increased costs, poorer prognosis, and higher mortality rates. However, there is currently no uniform definition or diagnostic criteria for frailty in stroke patients, and there is a need for standardized frailty assessments in this patient population.

The aim of this study is to determine the prevalence of frailty in stroke patients at the Stroke Unit of the University Hospital Giessen and to analyze the associated characteristics and impacts on clinical outcomes. A multimodal frailty assessment will be conducted to capture a wide range of frailty features and investigate their significance. The study includes all stroke patients admitted to the certified stroke- unit of the University Hospital Giessen within a 3-month period. There are no inclusion criteria related to age, gender, or type of stroke.

The multimodal frailty assessment encompasses determining appropriate blood values (e.g., CRP, albumin), assessing muscle strength/mass through handheld dynamometry and sonographic muscle diameter, utilizing scores like the Clinical Frailty Scale (CFS) and the Groningen Frailty Indicator (GFI), evaluating nutritional status (BMI), collecting image-based frailty data (e.g., sarcopenia, cerebral white matter lesions, lacunar strokes, brain atrophy), and conducting suitable one-year follow-ups. Additionally, demographic and clinical data such as age, gender, type of stroke, and treatment details will be recorded.

The primary outcome is the prevalence of frailty among stroke patients. Secondary outcomes include the characteristics and impacts of frailty in stroke patients, including correlations between various frailty features and clinical outcomes such as length of hospital stay, mortality, and functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* treated at the certified stroke-unit of the Dpt. of Neurology, University Hospital Giessen
* diagnosis of ischemic (including transient ischemic attack) or hemorrhagic stroke

Exclusion Criteria:

* withdrawal of care within 24 hours after admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted with the diagnosis of acute stroke treated at the certified stroke-unit will be included. All patients who consent for participation are further eligible for the outcome assessment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of frailty in stroke patients | 30 days
  Percentage of patients with frailty treated for stroke compared to all patients admitted for stroke
Rate of good functional outcome | 12 months
  Percentage of patients achieving a score of 0 to 2 on the modified Rankin scale (higher values indicating worse outcome, ranging from 0, no deficit, to 6, death) at 12 months follow-up

SECONDARY OUTCOMES:
Patient reported outcome measures (PROM) | 12 months
  Health-related quality measured using the visual analogue scale (VAS) of the Euroquol EQ-5D-3L tool. Score ranging from 0 to 100, with higher values indicating better quality of life.
Functional impairment in activities of daily living | 12 months
  Impairment in activities of daily living measuring the score on the Barthel-Index (BI; ranging from 0 to 100, with higher values indicating less impairment in activities of daily living).
Mortality rate | From date of admission until death or last follow-up, whichever comes first, assessed up to 12 months.
  Rate of death observed during the follow-up period
Cognitive outcome | 12 months
  Assessment of cognition using the telephone Montreal Cognitive Assessment test (tMOCA; ranging from 0 to 22, with a score of 18 or below indicating mild cognitive dysfunction)
Rate of rehospitalization | 12 months
  Percentage of patients needed to be hospitalized due to unplanned events during the follow-up
Major adverse cardiovascular events (MACE) | From date of admission until MACE or last follow-up, whichever comes first, assessed up to 12 months.
  Rate of patients suffering from newly detected myocardial infarction, non-fatal stroke or cardiovascular death

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Gerner, MD, Principal Investigator — Department of Neurology, University Hospital Giessen/Germany; Thorsten Doeppner, MD, Study Chair — Department of Neurology, University Hospital Giessen/Germany; Hagen Huttner, MD, PhD, Study Chair — Department of Neurology, University Hospital Giessen/Germany
Locations (1):
- Department of Neurology, University Hospital Giessen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Reasonable requests can be sent by mail.

REFERENCES:
- [Background] Giede-Jeppe A, Bobinger T, Gerner ST, Sembill JA, Sprugel MI, Beuscher VD, Lucking H, Hoelter P, Kuramatsu JB, Huttner HB. Neutrophil-to-Lymphocyte Ratio Is an Independent Predictor for In-Hospital Mortality in Spontaneous Intracerebral Hemorrhage. Cerebrovasc Dis. 2017;44(1-2):26-34. doi: 10.1159/000468996. Epub 2017 Apr 19. PMID 28419988
- [Background] Giede-Jeppe A, Reichl J, Sprugel MI, Lucking H, Hoelter P, Eyupoglu IY, Kuramatsu JB, Huttner HB, Gerner ST. Neutrophil-to-lymphocyte ratio as an independent predictor for unfavorable functional outcome in aneurysmal subarachnoid hemorrhage. J Neurosurg. 2019 Feb 1;132(2):400-407. doi: 10.3171/2018.9.JNS181975. Print 2020 Feb 1. PMID 30717052
- [Background] Gerner ST, Reichl J, Custal C, Brandner S, Eyupoglu IY, Lucking H, Holter P, Kallmunzer B, Huttner HB. Long-Term Complications and Influence on Outcome in Patients Surviving Spontaneous Subarachnoid Hemorrhage. Cerebrovasc Dis. 2020;49(3):307-315. doi: 10.1159/000508577. Epub 2020 Jul 3. PMID 32623428
- See also: website of the recruiting site: Dpt. of Neurology, University Hospital Giessen — https://www.ukgm.de/ugm_2/deu/ugi_neu/index.html